CLINICAL TRIAL: NCT02934425
Title: A Randomized, Controlled, Crossover Trial to Assess the Effects of a Lean Pork-containing, High-protein Breakfast on Indices of Satiety and Metabolic Health in Men and Women With Pre-diabetes
Brief Title: Effects of Lean Pork, High Protein Breakfast on Satiety and Metabolic Health in Pre-diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Midwest Center for Metabolic and Cardiovascular Research (Other)
Collaborators: National Pork Board (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: MC-1601
Record Dates: First submitted 2016-10-13; First posted 2016-10-17 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Pre-diabetes
Keywords: Pork; Refined carbohydrates; Satiety; Glucose; Insulin; Breakfast; Lipoprotein lipids
MeSH Terms: conditions — Glucose Intolerance; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Refined carbohydrate-rich breakfast (Placebo Comparator): Refined carbohydrate-rich breakfast
  Interventions: Other: Refined carbohydrate-rich breakfast
- High pork protein breakfast (Experimental): High pork protein breakfast
  Interventions: Other: High pork protein breakfast

INTERVENTIONS:
Other: Refined carbohydrate-rich breakfast — Refined carbohydrate-rich breakfast containing approximately 8/66/26% kcal from protein/carbohydrate/fat, respectively
  Arms: Refined carbohydrate-rich breakfast
Other: High pork protein breakfast — High pork protein breakfast containing approximately 35/39/26% kcal from protein/carbohydrate/fat, respectively
  Arms: High pork protein breakfast

SUMMARY:
The goal of this study is to assess the effects of consumption of a lean pork-containing, high-protein breakfast versus a refined carbohydrate-rich breakfast on satiety and cardiometabolic parameters in overweight or obese adults with pre-diabetes.

DETAILED DESCRIPTION:
This is a randomized, crossover trial that includes two screening visits, one baseline visit, and two test periods of 2 weeks each, each ending with a test visit, separated by a 2-week washout. Subjects consume each day a refined carbohydrate-rich breakfast containing 8/66/26% kcal from protein/carbohydrate/fat, respectively (Control Condition), or a high pork protein breakfast containing 35/39/26% kcal from protein/carbohydrate/fat, respectively (Active Condition). Study products for daily breakfast consumption will be dispensed to the subjects at the beginning of each test period. Subjects will complete 3-day diet records at baseline and the end of each test period, and a daily Appetite Visual Analog Scale (VAS) Diary to asses perceived hunger and fullness each evening before retiring throughout each test period. VAS assessments of hunger, fullness, desire to eat, prospective food consumption, focus and energy will also be assessed at the clinic visit at the end of each test period, pre- and post-breakfast consumption (multiple time points). Subjects will also complete a palatability questionnaire at the each of each test period. Blood samples will be collected at fasting at baseline and pre- and post-breakfast consumption (multiple sampling) at the end of each test period to evaluate glucose, insulin, and lipoprotein lipid concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index 25.0-39.9 kg/m2
* At least 1 of the following: a) capillary glycated hemoglobin 5.7-6.4%, b) fasting capillary glucose 100-125 mg/dL, or c) capillary glycated hemoglobin <5.7% and borderline fasting capillary glucose level 95-99 mg/dL and a subsequent fasting venous plasma glucose 100-125 mg/dL
* Self-identified "regular breakfast consumer" and willing to eat study foods as a breakfast meal
* Access to freezer and a food re-heating appliance
* Judged to be in good health on basis of medical history

Exclusion Criteria:

* Fasting laboratory test results of clinical significance (e.g., triglycerides ≥500 mg/dL, capillary glucose ≥126 mg/dL, glycated hemoglobin ≥6.5%)
* Uncontrolled hypertension
* Recent major trauma or surgical event
* Recent weight change ≥4.5 kg
* History or presence of clinically important endocrine, cardiovascular, pulmonary, biliary, or gastrointestinal disorders
* Recent history or presence of cancer (except non-melanoma skin cancer)
* History of extreme dietary habits
* Vegan or vegetarian
* History of eating disorder diagnosed by health professional
* Known intolerance or sensitivity to study products
* Unstable use of medications intended to alter lipid profile (e.g., unstable use of statins, bile acid sequestrants, cholesterol absorption inhibitor, fibrates, niacin-drug form, or omega-3-acid ethyl ester drugs)
* Recent use of foods or dietary supplements that might alter lipid metabolism (e.g., omega-3 fatty acid supplements or fortified foods, sterol/stanol products, pantethine, viscous dietary fiber supplements, red yeast supplements, garlic supplements, soy isoflavone supplements, probiotic supplements, niacin or analogues at >200 mg/d)
* Recent use of medications known to influence carbohydrate metabolism (e.g., adrenergic blockers, diuretics, hypoglycemic medications, systemic corticosteroids)
* Recent use of weight-loss drugs (including over-the-counter) or programs
* Recent history or current use of supplements and/or medications known to influence, satiety, appetite, taste, sense of smell, or weight (e.g., hypoglycemic medications and systemic corticosteroids)
* Recent use of antibiotics
* Signs or symptoms of active infection of clinical relevance
* Current or recent history of drug or alcohol abuse
* Pregnant, planning to be pregnant, or lactating females or women of childbearing potential unwilling to commit to use of a medically approved form of contraception

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-08; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Net incremental area under the curve (AUC) appetite VAS ratings | 2 weeks
  Difference between test conditions in net incremental AUC from pre-consumption (t = -15 minutes) to t = 240 minutes for VAS ratings for appetite (fullness, hunger, desire to eat, prospective food consumption)

SECONDARY OUTCOMES:
Net incremental AUC focus and energy VAS ratings | 2 weeks
  Difference between test conditions in net incremental AUC from pre-consumption (t = -15 minutes) to t = 240 minutes for VAS ratings for focus and energy
Total AUC VAS ratings | 2 weeks
  Difference between test conditions in total AUC from pre-consumption (t = -15 minutes) to t = 240 minutes for VAS ratings for appetite, focus and energy
Individual time points for VAS ratings | 2 weeks
  Difference between test conditions in fullness, hunger, desire to eat, prospective food consumption, and focus at individual time points from t = -15 minutes to t = 240 minutes
Energy intake at lunch | 2 weeks
  Difference between test conditions in the energy intake (kcal) at the lunch meal served at t = 240 minutes at the clinic visit at the end of each test period
Glucose total AUC and incremental AUC | 2 weeks
  Difference between test conditions in glucose total AUC and incremental AUC from 0 to 120 minutes and 0 to 240 minutes (the t = -15 minutes time point will be counted as t = 0 for this calculation)
Insulin total AUC and incremental AUC | 2 weeks
  Difference between test conditions in insulin total AUC and incremental AUC from 0 to 120 minutes and 0 to 240 minutes (the t = -15 minutes time point will be counted as t = 0 for this calculation)
Homeostasis model assessment of insulin sensitivity (HOMA-%S) | 2 weeks
  Difference between test conditions in HOMA-%S calculated from glucose and insulin values in samples collected at the end of each test period
Homeostasis model assessment of pancreatic beta-cell function (HOMA-%B) | 2 weeks
  Difference between test conditions in HOMA-%B calculated from glucose and insulin values in samples collected at the end of each test period
Lipoprotein lipids | 2 weeks
  Difference between test conditions in percent changes from baseline (day 0) to the end of each test condition (days 14 and 42) in triglycerides, total cholesterol, high-density lipoprotein cholesterol, low-density lipoprotein cholesterol, and non-high-density lipoprotein cholesterol
Triglyceride postprandial total AUC and incremental AUC | 2 weeks
  Difference between test conditions in postprandial total AUC and incremental AUC for triglycerides from 0 to 120 minutes and 0 to 240 minutes (the t = -15 minutes time point will be counted as t = 0 for this calculation)
Composite daily hunger and fullness VAS ratings | 2 weeks
  Difference between test conditions in the composite hunger and fullness VAS ratings from the daily Appetite VAS Dairy

CONTACTS AND LOCATIONS:
Overall Officials: Indika Edirisinghe, PhD, Principal Investigator — Illinois Institute of Technology; Kevin C Maki, PhD, Study Director — Midwest Center for Metabolic and Cardiovascular Research
Locations (1):
- Illinois Institute of Technology - Institute for Food Safety and Health, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No